CLINICAL TRIAL: NCT04863989
Title: Emergency Small vs Large Tube Thoracostomy in Chest Trauma Patients.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amr Mohamed Mamdouh Hussein, resident, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: small sized thoracostomy
Record Dates: First submitted 2020-09-17; First posted 2021-04-28 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Traumatic Pneumothorax and Hemothorax
MeSH Terms: conditions — Hemothorax

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Small sized chest tube (Experimental): Insertion of small sized chest tube in patients with traumatic hemothorax, pneumothorax or hemopneumothorax.
  Interventions: Procedure: tube thoracostomy
- Large sized chest tube (Active Comparator): insertion of large sized chest tube in patients with traumatic hemothorax, pneumothorax or hemopneumothorax.
  Interventions: Procedure: tube thoracostomy

INTERVENTIONS:
Procedure: tube thoracostomy — insertion of intercostal tube for drainage of traumatic hemothorax or pneumothorax

SUMMARY:
To compare between small sized tube thoracostomy and large sized tube thoracostomy regarding the need for another chest tube for the fear of obstruction (in hemomothorax) or ineffective drainage (in hemothorax, pneumothorax or hemo-pneumothorax) ,pain score or repositioning and need for thoracotomy.

DETAILED DESCRIPTION:
To evacuate abnormal fluid and air, chest tubes are placed in the pleural space, either surgically or percutaneously. Therapeutic drainage of pleural conditions such as pneumothorax, hemothorax, empyema, chylothorax, and malignant effusions, as well as prophylaxis drainage of air, blood, and other fluids after chest surgery are the indications for chest tubes.

Closed water-seal chest drainage has been described in 1875 by Gotthard Bülau to treat an empyema, as an alternative to the standard rib resection and open tube drainage in the acute phase or rib excision (saucerization) in the chronic phase.

Bülau emphasized the necessity of negative intrapleural pressure for re-expansion of a collapsed lung in the setting of thoracic empyema although most surgeons in his time attributed deaths from thoracic empyema to infection and not superimposed respiratory compromise due to open pneumothorax .

He understood that closed water seal drainage could facilitate lung re-expansion via the patient's natural respiratory movements. Unfortunately, until mechanical ventilation was introduced, application of these principles was limited to the treatment of thoracic empyema.

During both the Second World War and the Korean one lung function restoration was the primary goal of thoracic wound treatment: emergency tube thoracostomy became extremely frequent in haemothorax and tension pneumothorax treatment. For the first time the drain was connected to a two-bottle water seal suction system since 1952 , synthetic ones, more flexible and easy to place, replaced metal tubes and modern three chamber thoracic drain, for a more efficient suction, were employed. New, flexible and plastic drains were widely used by the 1980s, they ranged between 6 and 40 French (F) in size. Since it was believed that smaller drains were less effective in adult medicine, being more prone to the risk of obstruction, the smaller ones (≤20 F) were commonly used in children, the bigger in adults,. In the last two decades, small-bore chest tubes (SBCT) have gained increasing popularity In traumatic pneumothorax or hemothorax the optimal tube size for an emergent thoracostomy is unknown. For the nonemergent management of patients with traumatic pneumothorax or hemothorax both small catheter tube thoracostomy and large-bore chest tube thoracostomy have been shown to work.

In stable trauma patients small catheter tube thoracostomy is effective and comparable with large catheter tube thoracostomy in managing chest trauma.

While the available evidence suggests that in resolving traumatic haemothoraces without additional complications small bore drains may be as effective as large bore drains, there is insufficient evidence currently available to recommend a change to standard practice (ie, large bore drains).

Inaba K , et al, 2012 concluded that chest tube size did not impact the clinically relevant outcomes tested for injured patients with chest trauma. There was no difference in the efficacy of drainage, need for additional tube drainage, or invasive procedures and rate of complications including retained hemothorax. Pain felt by patients at the site of insertion was not affected by tube size.

Most occurrences of traumatic pneumothorax (PTX) and hemothorax (HTX) can be managed non-operatively by means of chest tube thoracostomy. Although most guidelines for chest trauma recommend a large-bore chest tube, e.g., the 9th edition of the ATLSTM (Advanced Trauma Life Support) program recommends a 36 or 40 Fr tube, and the JATECTM (Japan Advanced Trauma Evaluation and Care) course recommends a 28 Fr or larger tube and choosing the tube size based on the patient's physique, these recommendations are mainly based on traditional clinical habits. These large-bore chest tubes may cause pain related to the insertion site and discomfort, especially in conscious patients. Smaller tubes were reported to reduce the pain associated with the tube insertion site in patients with pleural infection.

ELIGIBILITY:
Inclusion Criteria:

* all chest trauma patients with significant hemothorax, pneumothorax or combined hemo-pneumothorax

Exclusion Criteria:

* any chest trauma patients undergoing thoracotomy or thoracic surgery for any other reason for example : diaphragmatic tear,flail chest or sternal fracture

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
To compare the number of patients who will have emergent small sized tube thoracostomy and large sized tube thoracostomy regarding the need for another chest tube. | baseline
  To compare the number of patients who will have emergent small sized tube thoracostomy and large sized tube thoracostomy regarding the need for another chest tube.

SECONDARY OUTCOMES:
Number of trauma patients who will have emergent small vs large thoracostomy tube regarding pain score | baseline
  Number of trauma patients who will have emergent small vs large thoracostomy tube regarding pain score
Number of trauma patients who will have emergent small vs large thoracostomy tube regarding duration of tube insertion. | baseline
  Number of trauma patients who will have emergent small vs large thoracostomy tube regarding duration of tube insertion.

REFERENCES:
- [Background] Cooke DT, David EA. Large-bore and small-bore chest tubes: types, function, and placement. Thorac Surg Clin. 2013 Feb;23(1):17-24, v. doi: 10.1016/j.thorsurg.2012.10.006. PMID 23206714
- [Background] Meyer JA. Gotthard Bulau and closed water-seal drainage for empyema, 1875-1891. Ann Thorac Surg. 1989 Oct;48(4):597-9. doi: 10.1016/s0003-4975(10)66876-2. PMID 2679468
- [Background] Van Schil PE. Thoracic drainage and the contribution of Gotthard Bulau. Ann Thorac Surg. 1997 Dec;64(6):1876. No abstract available. PMID 9436605
- [Background] Monaghan SF, Swan KG. Tube thoracostomy: the struggle to the "standard of care". Ann Thorac Surg. 2008 Dec;86(6):2019-22. doi: 10.1016/j.athoracsur.2008.08.006. PMID 19022041
- [Background] HOWE BE Jr. Evaluation of chest suction with an artificial thorax. Surg Forum. 1951:1-7. No abstract available. PMID 14931188
- [Background] Miller KS, Sahn SA. Chest tubes. Indications, technique, management and complications. Chest. 1987 Feb;91(2):258-64. doi: 10.1378/chest.91.2.258. No abstract available. PMID 3542404
- [Background] Filosso PL, Sandri A, Guerrera F, Ferraris A, Marchisio F, Bora G, Costardi L, Solidoro P, Ruffini E, Oliaro A. When size matters: changing opinion in the management of pleural space-the rise of small-bore pleural catheters. J Thorac Dis. 2016 Jul;8(7):E503-10. doi: 10.21037/jtd.2016.06.25. PMID 27499983
- [Background] Tanizaki S, Maeda S, Sera M, Nagai H, Hayashi M, Azuma H, Kano KI, Watanabe H, Ishida H. Small tube thoracostomy (20-22 Fr) in emergent management of chest trauma. Injury. 2017 Sep;48(9):1884-1887. doi: 10.1016/j.injury.2017.06.021. Epub 2017 Jun 23. PMID 28673640
- [Background] Rivera L, O'Reilly EB, Sise MJ, Norton VC, Sise CB, Sack DI, Swanson SM, Iman RB, Paci GM, Antevil JL. Small catheter tube thoracostomy: effective in managing chest trauma in stable patients. J Trauma. 2009 Feb;66(2):393-9. doi: 10.1097/TA.0b013e318173f81e. PMID 19204512
- [Background] Towards evidence-based emergency medicine: best BETs from the Manchester Royal Infirmary. BET 4: does size matter? Chest drains in haemothorax following trauma. Emerg Med J. 2013 Nov;30(11):965-7. doi: 10.1136/emermed-2013-203139.4. PMID 24142946
- [Background] Inaba K, Lustenberger T, Recinos G, Georgiou C, Velmahos GC, Brown C, Salim A, Demetriades D, Rhee P. Does size matter? A prospective analysis of 28-32 versus 36-40 French chest tube size in trauma. J Trauma Acute Care Surg. 2012 Feb;72(2):422-7. doi: 10.1097/TA.0b013e3182452444. PMID 22327984
- [Background] ATLS Subcommittee; American College of Surgeons' Committee on Trauma; International ATLS working group. Advanced trauma life support (ATLS(R)): the ninth edition. J Trauma Acute Care Surg. 2013 May;74(5):1363-6. doi: 10.1097/TA.0b013e31828b82f5. No abstract available. PMID 23609291